CLINICAL TRIAL: NCT00260767
Title: An Imaging Trial of the Distribution of Topical Gel in the Human Vagina: Enhanced MRI Techniques to Increase Resolution
Brief Title: Imaging Trial of the Distribution of Topical Gel in the Human Vagina: Enhanced MRI Techniques to Increase Resolution
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Biosyn (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRU009
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2005-12-02 (Estimated); Status verified 2005-11

CONDITIONS: HIV

INTERVENTIONS:
Drug: HEC placebo gel

SUMMARY:
This study will assess the distribution of topical gel in the human vagina, using enhanced MRI techniques. The number and size of uncovered areas will be studied, and the upper genital tract will be examined for the presence of topical gel using MRI.

DETAILED DESCRIPTION:
This study will assess the distribution of topical gel in the human vagina, using enhanced MRI techniques. The number and size of uncovered areas will be studied, and the upper genital tract will be examined for the presence of topical gel using MRI. MRIs will be performed with both a standard pelvic coil and an enhanced resolution endo-rectal coil in order to obtain maximal resolution. MRI images will be acquired before and after simulated coitus.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 year old women
* not pregnant
* willingness to use effective method of contraception
* regular menstrual cycle
* normal Pap test result

Exclusion Criteria:

* abnormal pelvic exam
* pregnant or breastfeeding
* claustrophobia or other MRI contraindications
* hypertension, hemolytic anemia,latex allergy
* history of hemorrhoids or irritable bowel syndrome

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6

PRIMARY OUTCOMES:
1. Number and size of bare spots, before and after simulated coitus.
2. Number of women with migration of gel into the endocervical canal and/or endometrial canal before and after simulated coitus.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Barnhart, MD, Principal Investigator — University of Pennsylvania Medical Center
Locations (1):
- Reproductive Research Unit, U of Penn Medical Center, Philadelphia, Pennsylvania, United States